CLINICAL TRIAL: NCT02450617
Title: Stabilizing Group Treatment of Complex Trauma: A Randomized Controlled Trial
Acronym: STAB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Modum Bad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Oslo
Record Dates: First submitted 2015-05-13; First posted 2015-05-21 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Posttraumatic Stress Disorder; Dissociative Identity Disorder; Dissociative Disorder
Keywords: Complex PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Dissociative Identity Disorder; Dissociative Disorders | interventions — Coping Skills

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Stabilizing group treatment for PTSD (Experimental): Group treatment, 20 sessions psychoeducation and skills-training. In combination with conventional individual treatment.
  Interventions: Behavioral: Conventional individual treatment; Behavioral: Stabilizing group treatment for PTSD
- Conventional Individual treatment - PTSD (Active Comparator): Conventional individual treatment.
  Interventions: Behavioral: Conventional individual treatment
- Stabilizing group treatment for Dissociative disorders (Experimental): Group treatment, 20 sessions psychoeducation and skills-training. In combination with conventional individual treatment.
  Interventions: Behavioral: Conventional individual treatment; Behavioral: Stabilizing group treatment for Dissociative disorders
- Conventional Individual treatment - Dissociative disorders (Active Comparator): Conventional individual treatment.
  Interventions: Behavioral: Conventional individual treatment

INTERVENTIONS:
Behavioral: Conventional individual treatment — Individual psychotherapeutic treatment and case-management delivered by public outpatient clinics or private practicing psychologist/psychiatrist
Behavioral: Stabilizing group treatment for PTSD — 20 sessions group psychotherapy for patients with PTSD, focused on psychoeducation and skills-training.
  Other Names: "Back to here and now"
  Arms: Stabilizing group treatment for PTSD
Behavioral: Stabilizing group treatment for Dissociative disorders — 20 sessions group psychotherapy for patients with PTSD, focused on psychoeducation and skills-training
  Other Names: "Coping with Trauma-Related Dissociation"
  Arms: Stabilizing group treatment for Dissociative disorders

SUMMARY:
The research project outlined in this proposal aims to investigate the effectiveness of stabilizing group treatment as an add-on to conventional treatment, for patients with Post Traumatic Stress Disorder (PTSD) or dissociative disorders after childhood abuse. The investigators also aim to study psychophysiological markers associated with complex trauma and treatment, mechanisms of change involved in treatment, and which patient characteristics that predict positive outcome.

DETAILED DESCRIPTION:
Patients with histories of repeated traumatization in childhood often display a wide array of symptoms described as complex traumatic stress disorder. This sequela involves a high degree of comorbid mental and somatic disturbances, and entails tremendous health care costs for society and suffering for the victims. Despite the prevalence and consequences of complex trauma, research on effective treatments is extremely limited. Expert clinicians suggest that initial treatment for these patients should focus on stabilization of symptoms through psychoeducation and skills - training, and some research has supported this advice. Offering such treatment as group therapy can be both cost - effective and give patients additional peer-support. The research project outlined in this proposal aims to investigate the effectiveness of stabilizing group treatment as an add-on to conventional treatment, for patients with PTSD or dissociative disorders after childhood abuse. This will be investigated in a randomized controlled design. The investigators also aim to discover psychophysiological markers associated with treatment, mechanisms of change involved in treatment, and what patient characteristics that predict outcome. The results may contribute to new knowledge about treatment of complex traumatization, as well as new and improved health services for a vulnerable patient group with little specialized treatment today.

The main aim of this project is to compare the effectiveness of stabilizing group treatment as an add-on to conventional individual therapy, to conventional individual therapy alone, in a randomized controlled design. This will be tested in two independent diagnostic groups: Patients with PTSD and patients with Dissociative disorders, both groups with reports of childhood abuse. The investigators will further investigate how level of dissociative symptoms influence treatment, how group climate influence symptoms, the relationship between individual and group therapy in combined treatment, and how treatment affects Heart Rate Variability. The investigators also seek to evaluate the treatment economically with a societal perspective, carrying out cost-utility analyses.

ELIGIBILITY:
* The inclusion criteria will be similar to clinical practice to ensure the external validity of the research.

  * participants must report a history of childhood abuse
  * be between 18 and 65 years of age
  * have enough competence in Norwegian to be able to participate in a psychoeducational group.
* In the PTSD arm of the study patients must meet the criteria for a DSM - 5 diagnosis of Posttraumatic Stress Disorder.
* In the Dissociative-disorders arm of the study the patients must meet criteria for a DSM-5 diagnosis of Dissociative Identity Disorder (DID) or Dissociative Disorder Not Otherwise Specified (DDNOS).

Exclusion criteria will include:

1. Acute suicidality
2. Serious substance abuse interfering with treatment
3. Serious psychotic symptoms
4. Current life - crisis interfering with therapy (e.g. ongoing abuse, divorce, court case, somatic disease in spouse or children, etc.)
5. Neurological disease, mental disability or life threatening somatic disease. For the PTSD arm of the study an additional exclusion criteria will be that the patient meets the criteria for a dissociative disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2014-06; Primary Completion 2019-09 (Actual); Study Completion 2019-09 (Actual)

PRIMARY OUTCOMES:
Global Assessment of Functioning - change from baseline | 1 week after completed treatment
  Daily life functioning and severity of symptoms last week, assessed by interview
Global Assessment of Functioning- change from baseline | 6 months after completed treatment
  Daily life functioning and severity of symptoms last week, assessed by interview

SECONDARY OUTCOMES:
Heart rate variability- change from baseline | 1 week after completed treatment
  Resting state heart rate variability
Heart rate variability - change from baseline | 6 months after completed treatment
  Resting state heart rate variability
PTSD Symptom Scale - Self-Report - change from baseline | 1 week after completed treatment
PTSD Symptom Scale - Self-Report - change from baseline | 6 months after completed treatment
Symptom Checklist 90 Revised - change from baseline | 1 week after completed treatment
Symptom Checklist 90 Revised - change from baseline | 6 months after completed treatment
Inventory of Interpersonal Problems - change from baseline | 1 week after completed treatment
Inventory of Interpersonal Problems - change from baseline | 6 months after completed treatment
Dissociative Experiences Scale II - change from baseline | 1 week after completed treatment
Dissociative Experiences Scale II - change from baseline | 6 months after completed treatment
Behavior Checklist - change from baseline | 1 week after completed treatment
  registers function and self-destructive behavior
Behavior Checklist - change from baseline | 6 months after completed treatment
  registers function and self-destructive behavior
Short Form 36 - change from baseline | 1 week after completed treatment
Short Form 36 - change from baseline | 6 months after completed treatment

OTHER OUTCOMES:
Use of health services - change from 6 months pre-treatment | 6 months after completed treatment
  Assessed by data from Norwegian Patient Register

CONTACTS AND LOCATIONS:
Locations (1):
- Traumepoliklinikken, Modum Bad i Oslo, Oslo, Norway

REFERENCES:
- [Derived] Baekkelund H, Ulvenes P, Boon-Langelaan S, Arnevik EA. Group treatment for complex dissociative disorders: a randomized clinical trial. BMC Psychiatry. 2022 May 16;22(1):338. doi: 10.1186/s12888-022-03970-8. PMID 35578194